CLINICAL TRIAL: NCT02492828
Title: Adherence of Apixaban and Warfarin in Patients With Atrial Fibrillation in Real-world Setting in Sweden
Brief Title: Adherence of Apixaban and Warfarin in Patients With Arterial Fibrillation in Real-world Setting in Sweden
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CV185-323
Record Dates: First submitted 2015-06-30; First posted 2015-07-09 (Estimated); Last update posted 2016-05-18 (Estimated); Status verified 2016-05

CONDITIONS: Anticoagulation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients for filled prescriptions for apixaban
- Patients for filled prescriptions for warfarin

SUMMARY:
This will be a retrospective cohort study using national register linkage data (including prescription, inpatient, mortality, and socioeconomic data). The study period will be from May 29, 2013 to June 30, 2015. Patients will be followed from the start of treatment (index date) until their death, exiting the database, or until the end of the study period (June 30, 2015).

ELIGIBILITY:
Inclusion Criteria:

* For the AF cohort

  * Patients that have ≥1 AF diagnosis registered in the patient register
* Apixaban subcohort 1

  * Patients eligible for the AF cohort
  * Patients that had a first prescription for apixaban during the identification period without previous prescriptions for NOACs or warfarin during the preceding 12 months
* Warfarin subcohort 1

  * Patients eligible for the AF cohort
  * Patients that had a first prescription for warfarin during the identification period without previous prescriptions for NOACs or warfarin during the preceding 12 months
* Apixaban subcohort 2

  * Patients eligible for the AF cohort
  * Patients that had a first prescription for apixaban during

Exclusion Criteria:

* For the AF cohort:

  * Patients with valvular AF will be excluded (see definition Appendix 1)
* Warfarin subcohort 1:

  * Patients will be excluded from this sub-cohort if they had at least one prescription for warfarin or NOACs during the 12-month period preceding the first prescription for warfarin during the identification period, ie, the index date

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will include all patients with filled prescriptions for apixaban or warfarin between May 29, 2013 and Dec 31, 2014 that are identified with a hospital diagnosis of non-valvular atrial fibrillation (NVAF)
Sampling Method: Non-Probability Sample
Enrollment: 41000 (Actual)
Dates: Start 2014-06; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Compare adherence among Atrial Fibrillation (AF) patients initiating treatment with apixaban (without previous warfarin or novel anticoagulant (NOAC) use) compared with those initiating treatment with warfarin (without previous warfarin or NOAC use) | approximately 6 to 12 months
  Adherence: Adherence will be defined including missing doses and treatment discontinuation using the following approaches:
  "Drug at disposal" approach: Based on information on prescribed dosing (mg/day) and information on filled prescriptions (mg expensed from the pharmacy); it is possible to calculate for how long a period the drug will last for that specific patient. Adherence is then defined using the Medication Possession Ratio (MPR) calculated as the ratio of number of days of treatment supply divided by the total length of follow-up time, and converted to a percentage (in the graph below illustrated as the sum of the grey horizontal bars divided by the length of follow-up, ie, time between index date and end of follow-up). The MPR will be computed as a continuous and binary variable (MPR>80%, ie, high vs low adherence)
Compare persistence among AF patients initiating treatment with apixaban (without previous warfarin or NOAC use) compared with those initiating treatment with warfarin (without previous warfarin or NOAC use) | approximately 6 to 12 months
  Persistence: Persistence will be defined as treatment discontinuation and will be measured by estimating the following:
  * Time to discontinuation: Date of therapy cessation is not possible to determine with certainty due to the nature of registry data. In order to be able to estimate the time of discontinuation, patients will be considered on treatment for the full time between two purchases as long as they have at least one refill in a six month period. If there is no new purchase within six months the patient is considered to have terminated treatment at a date corresponding to how long the last prescription will last (in the graph below illustrated as the time between index date and the end of the "last" horizontal bar).
  * Cumulative incidence of persistent patients still on index treatment at the every 3- month interval after index date (treatment initiation)

SECONDARY OUTCOMES:
Describe and compare patient characteristics (demographics) among AF patients through questionnaire | approximately 6 to 12 months
  Describe and compare patient characteristics (eg, demographics and clinical) among AF patients who:
  * Initiate apixaban without previous anticoagulant treatment (warfarin or NOAC use)
  * Initiate apixaban with previous war
  Demographic parameters : Age-groups, Sex, Socioeconomic variables (e.g. education, disposable income)
Describe and compare patient characteristics (clinical) among AF patients through questionnaire | approximately 6 to 12 months
  Describe and compare patient characteristics (eg, demographics and clinical) among AF patients who:
  * Initiate apixaban without previous anticoagulant treatment (warfarin or NOAC use)
  * Initiate apixaban with previous war
  Clinical Characteristics: History of stroke/TIA/systemic, embolism, Diabetes, Hypertension, Heart failure, Vascular disease, Intracranial bleeding, Any bleeding, Kidney disease, Liver disease, Dementia, Valvular AF, Ischemic stroke, Unspecified stroke, TIA, Systemic embolism, Coronary disease, End Stage Renal Disease

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb

REFERENCES:
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx